CLINICAL TRIAL: NCT03077334
Title: Oncologic Outcomes Based on Clinical Pattern of Preoperative PET-CT in Resected Pancreatic Cancer-Prospective Cohort Study
Brief Title: Oncologic Outcomes Based on Clinical Pattern of Preoperative PET-CT in Resected Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0702
Record Dates: First submitted 2017-02-20; First posted 2017-03-10 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- K-type: FDG uptake in pancreatic cancer is similar to that of kidney
  Interventions: Device: PET-CT
- non K-type: FDG uptake in pancreatic cancer is lower than that of kidney
  Interventions: Device: PET-CT

INTERVENTIONS:
Device: PET-CT — PET-CT will be done before operation and that is routine treatment procedure for pancreatic cancer.

SUMMARY:
The 18F-FDG-PET scan is currently being used for cancer diagnosis, staging, identifying hidden metastasis, and assessment of treatment responses in clinical oncology. Although there are important studies suggesting potential associations between PET-based parameters and oncologic outcomes, the calculation and official documentation of individual PET-based parameters might not be routine in clinical practice because these processes usually require time- and labor-consuming processes for the radiologists. In this study, the investigators prospectively determined clinical 18F-FDG-PET type according to degree of FDG-uptake in pancreatic cancer and compare oncologic outcomes between the types.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for radical pancreatectomy due to pancreatic cancer without neoadjuvant treatment
* Age between 20 years old and 80 years old
* General performance status greater than 70
* Results of peroperative PET-CT available

Exclusion Criteria:

* Unresectable, locally advance and metastatic pancreatic cancer
* Patients not wanting operation
* ASA score of greater than 3
* History of chronic alcoholism ot drug abuse
* Lack of patient compliance
* Patients not agreeing to enroll in the study.
* Patients unable to understand and sign the study agreement.
* History of neoadjuvant treatment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Referral Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Clinical PET type assessed by surgeons from preoperatively preformed PET imaging | 1 week after surgery
  Three surgeons will review the preoperative PET imaging and each will determine the clinical PET type as either K-type or Non-K type. Inter-surgeon agreement of clinical PET type will be determined. Clinicopathologic characteristics between K-type and Non-K type will also be analyzed.

SECONDARY OUTCOMES:
Number of patients with recurrence of cancer or mortality from cancer following operation | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepatobiliary and Pancreatic Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided